CLINICAL TRIAL: NCT07388537
Title: .]Yere Evaluation of the Clinical Spectrum of Diabetes and Obesity in Youth and Adults
Brief Title: Evaluation of the Clinical Spectrum of Diabetes and Obesity in Youth and Adults
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002229; 002229-DK
Record Dates: First submitted 2026-02-04; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Obesity; Diabetes; Metabolic Disorders
Keywords: Clinical Spectrum of Diabetes; Obesity; Hyperglycemia; Metabolic Disease
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Diseases; Hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults with suspected or established hyperglycemia, overweight or obesity, or metabolic disease: Data and samples will be obtained during complete comprehensive clinical screening procedures and provision of standard of care treatments. Data and samples to be retained may include either residual samples/ data not otherwise needed for clinical care or additional samples/ data collected during the course of clinical care. These data will provide information to prevent the development and/or progression of cardiovascular disease and other diabetes-related complications, to increase the understanding of these disease processes in patients with different age of onset of metabolic disease, and how available treatments affect the prognosis in these patients.
- Youth with suspected or established hyperglycemia, overweight or obesity, or metabolic disease: Data and samples will be obtained during complete comprehensive clinical screening procedures and provision of standard of care treatments. Data and samples to be retained may include either residual samples/ data not otherwise needed for clinical care or additional samples/ data collected during the course of clinical care. These data will provide information to prevent the development and/or progression of cardiovascular disease and other diabetes-related complications, to increase the understanding of these disease processes in patients with different age of onset of metabolic disease, and how available treatments affect the prognosis in these patients.

SUMMARY:
Background:

Diabetes and obesity are chronic diseases. They can affect blood flow and how the body processes nutrients, and complications over time can lead to early death. Diabetes can affect children as well as adults, but the disease seems to be more severe and to progress faster when it appears in younger people. Researchers want to understand more about how diabetes and obesity develop and change over time.

Objective:

To collect data and samples regularly from people with obesity and diabetes.

Eligibility:

People aged 8 to 65 years. They must be overweight or obese; or have high blood sugar; or have problems with how their body uses food for energy.

Design:

Participants will have additional procedures during routine care visits at the NIH clinic.

Data collected for the study will include the following:

Information from the participant s medical chart will be kept for research.

Questionnaires will ask about participant s eating habits, feelings, sleep, and substance use. They will take 30 to 60 minutes. Care providers will address any issues revealed in these surveys.

Blood, saliva, urine, and stool samples will be collected. Samples may be used for genetic tests.

Data and samples will be kept for future research.

Participants may remain in the study up to 30 years.

DETAILED DESCRIPTION:
Study Description:

This is a single-site observational study conducted at the NIH Clinical Center. Youth and adults who have suspected or established hyperglycemia, overweight or obesity, or metabolic disease, or who require clinical screening for such conditions are provided standard clinical care. Data and samples obtained during regular clinical care will be retained for future research. Recommendations for other treatment options outside of the NIH will be discussed with study participants and may be discussed with their primary or referring physicians.

The schedule a participant follows will be based on their unique clinical needs.

Objectives:

To collect data and samples during clinical evaluation, treatment, and follow-up of participants for use in future studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age 8 years to 65 years
2. Meet at least one of the following:

   a. Overweight/Obesity:

   i. For participants under 18 years of age: BMI >= 85th percentile for age and sex

ii. For participants >= 18 years of age: BMI >= 25 kg/m^2 (>=23 kg/m^2 for self-reported Asian race/ethnicity)

b. Suspected or evidence of hyperglycemia:

i. Diagnosis of prediabetes or diabetes in medical history or by participant/guardian/Legally Authorized Representative (LAR) report, OR

ii. Fasting blood glucose >= 100 mg/dL in medical record, OR

iii. Postprandial blood sugar >= 140 mg/dL in medical record, OR

iv. Hemoglobin A1c >= 5.7% in medical record

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of significant medical illnesses that the investigators feel may interfere with potential evaluations, i.e. individuals who are critically ill, unstable, or with severe organ failure that may affect/limit the endocrine evaluation and place unsustainable demands on Clinical Center or NIDDK resources.
2. History of any medical, psychiatric, or social conditions which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the participant.
3. Inability or unwillingness of participant, parent/guardian, or LAR to provide informed consent.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a single-site observational study conducted at the NIH Clinical Center. Youth and adults who have suspected or established hyperglycemia, overweight or obesity, or metabolic disease, or who require clinical screening for such conditions are provided standard clinical care. Data and samples obtained during regular clinical care will be retained for future research. Recommendations for other treatment options outside of the NIH will be discussed with study participants and may be discussed with their primary or referring physicians. The schedule a participant follows will be based on their unique clinical needs.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2054-11-30 (Estimated); Study Completion 2055-04-30 (Estimated)

PRIMARY OUTCOMES:
To collect data and samples during clinical evaluation, treatment, and follow-up of participants for use in future studies. | Up to 30 years
  Samples including whole blood, saliva/buccal swabs, urine, and/or stool will be collected and stored for use in future studies to test our hypothesis that individuals with youth and adult early-onset diabetes and obesity will have high rates of metabolic complications and rapid disease progression compared to adults who develop diabetes later in their life. These samples will be collected during the participants' clinical care visits

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Malandrino, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
For associate protocols, identifiable data will be de-identified prior to repository submission. Participant level clinical data related to primary outcomes, will be preserved through deposition of the data in a controlled access public repository.
Supporting Information: Study Protocol
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscript will be available at the time of publication. All other generated data will be shared no later than at the end of the award.
Access Criteria: The study protocol, data dictionary and a glossary of domain-specific terms to facilitate interpretation of scientific data related to primary outcomes will be submitted.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002229-DK.html